CLINICAL TRIAL: NCT07151248
Title: ELECTRIG: Evaluating Effects of Cranial Electrical Stimulation Therapy With Responsive Imaging in Gulf War Illness Pain and Comorbid Symptoms
Brief Title: Cranial Electrotherapy Stimulation and Brain Imaging for Gulf War Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anna Woodbury, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00009810; GRANT14297332 (Other Grant/Funding Number: Department of Defense); GRANT14297241 (Other Grant/Funding Number: Department of Defense); 2025P011630 (Other: Emory IRB)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gulf War Syndrome
Keywords: Gulf War Illness Headaches and Pain
MeSH Terms: conditions — Persian Gulf Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, sham-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- True CES therapy (Experimental): The participant will be trained in device usage and instructed to use the device each evening around the same time for 60 minutes (timer will be pre-set). The intervention (true CES) will occur over the course of 6 weeks.
  Interventions: Device: Cranial electrical/electrotherapy stimulation (CES)
- Sham CES therapy (Sham Comparator): The participant will be trained in device usage and instructed to use the device each evening around the same time for 60 minutes (timer will be pre-set). The intervention (sham CES) will occur over the course of 6 weeks.
  Interventions: Device: Sham Cranial electrical/electrotherapy stimulation (CES)
- True CES therapy for non-responders (Experimental): For the non-responders (<2 point decrease on DVPRS), the blind will be broken, and those non-responder participants who were initially assigned to sham placebo CES during the first 6 weeks of the intervention, now will be offered the opportunity to utilize the true CES device in a modified sequential parallel comparison design for an additional 6 weeks.
  Interventions: Device: Cranial electrical/electrotherapy stimulation (CES)

INTERVENTIONS:
Device: Cranial electrical/electrotherapy stimulation (CES) — Cranial electrical/electrotherapy stimulation (CES) is a non-pharmacological, portable, non-invasive intervention.
  Active research units will be locked at the specified amplitude and administer that amplitude of stimulation for 60 minutes therapy.
  Other Names: CES, Alpha-Stim™
  Arms: True CES therapy; True CES therapy for non-responders
Device: Sham Cranial electrical/electrotherapy stimulation (CES) — Sham research units will be locked into active sham mode which provides stimulation designed to provide the sensation of stimulation for only 5 minutes while continuing to count down for the remaining 55 minutes.
  Arms: Sham CES therapy

SUMMARY:
The main goal of the proposed study is to critically evaluate a nonpharmacological and readily available therapy, cranial electrical stimulation (CES) using Alpha-Stim™, and to discover the brain function mechanisms underlying Gulf War Illness-related Headache and Pain (GWI-HAP) and treatment response to CES.

For this objective, the investigators will employ an adaptive trial design as well as a neuroimaging technique using MRI, which has become the pre-eminent technique for assessing the integrity of brain function, connectivity, and organization in healthy brain and pathology.

DETAILED DESCRIPTION:
Gulf War Veterans are disproportionately plagued by fibromyalgia-like symptoms including headaches, joint, and muscle pain, known as gulf war illness pain or GWI-HAP. Treatment options are limited, and the neurobiology of these symptoms is poorly understood.

In this population, the investigators plan to test a portable, non-pharmacological, non-invasive therapy (Alpha-Stim™) that is FDA-cleared for anxiety, insomnia, and pain, and readily available for widespread implementation in the United States. This cranial electrical stimulation (CES) device has shown promising, though limited results for anxiety, insomnia, and pain. They also plan to employ magnetic resonance spectroscopy (MRS) to evaluate neuroinflammation.

Subjects will be male and females, age 40-80 years old, with a diagnosis of Gulf war illness. Subjects will be recruited by referral and posted flyers on Emory campus, ResearchMatch, the Gulf War Registry, and the Wounded Warriors' Program. The research team will not approach vulnerable populations including minors, prisoners, pregnant persons, neonates or human fetuses, wards of the state, or cognitively impaired persons. Recruitment, screening and enrollment will occur at the Emory clinics (EUHM and EUH) and the Human Subjects Research Building II.

This randomized, double-blind, sham-controlled study will compare the efficacy of "active" or true CES therapy to "sham" CES therapy. Participants will be randomized in a 1:1 ratio to true or sham CES (n=104 total; 52 true, 52 sham). Up to 130 subjects will be enrolled to achieve 104 treated subjects. Baseline assessments including quality of life questionnaires and pain assessments, in addition to MRI will be obtained prior to initiation of the intervention.

The participant will be trained in device usage and instructed to use the device each evening around the same time for 60 minutes (timer will be pre-set). They will also be provided detailed instructions.

The intervention (both sham and true CES) will occur over the course of 6 weeks, and participants will be assessed again post-treatment. To assess our neuroimaging outcomes, MRI will also be obtained at 6 weeks post-treatment, to assess for changes in connectivity and neuroinflammation. The total time commitment for most subjects will be 7 weeks.

Participants who are initially randomized to sham and are determined to be non-responders (<2 point decrease on DVPRS) will be offered the opportunity to utilize the true CES therapy with additional reimbursement and follow-up periods. They will use the device for an additional 6 weeks and return for post-treatment follow up at that time (12 weeks after initial therapy) that will include additional MRI and the original baseline and 6-week assessments. The total time commitment for these subjects will be 13 weeks.

A verbal prescreening consent will be used to confirm eligibility. Informed consent will be conducted in person with the participant and written, or over the telephone or zoom with consent signed using Hipaa Part 11 compliant DocuSign. Participants may also consent to be contacted for future research.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male and female age 40-80 years old
2. Meet criteria for GWVI based on the CDC and Kansas Criteria for GWVI.

   * CDC: 1 or more from at least 2 of the following categories for ≥ 6 months): 1) fatigue 2) mood and cognition (symptoms of feeling depressed, difficulty in remembering or concentrating, feeling moody, feeling anxious, trouble in finding words, or difficulty in sleeping) 3) musculoskeletal (symptoms of joint pain, joint stiffness, or muscle pain
   * Kansas: 3 of 6 domains: 1) fatigue and sleep problems 2) pain symptoms 3) neurologic, cognitive, or mood symptoms 4) gastrointestinal symptoms 5) respiratory symptoms 6) skin symptoms chronic since 1990. Symptom reporting must be in the absence of diagnosed exclusionary conditions; only respondents who have at least 1 moderately severe symptom or 2 or more symptoms within a group were considered to have a high level of symptoms in the group.
3. Subjects must self-report consistent, daily pain (greater than or equal to 4 on the DVPRS) >90 days (prior to enrollment)
4. Subjects must have intact skin free of infection at the site of electrode placement (earlobe).
5. Subjects must be willing to participate and understand the consent.
6. Subjects must be right-handed to provide consistency in brain structure and function.

Exclusion Criteria:

1. Subjects must not be currently pregnant since effects of fMRI and electrical current on the developing fetus are not well-known.
2. Subjects must not have a history of drug abuse or severe, uncontrolled psychiatric illness such as schizophrenia or major depressive disorder with suicidal ideation.
3. Subjects must not have psoriasis vulgaris or other skin conditions that may increase the risk of infection at the implantation site.
4. Subjects must not introduce new medications or treatments for symptoms during the study to prevent confounding results.
5. Subjects must not have severe anxiety, claustrophobia, or other conditions that may prevent their ability to lie at rest in an MRI scanner. This will be determined after discussion with the patient regarding their own perceived ability to lie at rest in an MRI scanner without the use of additional sedating medications.
6. Subjects must not have an implanted electrical device such as a surgically placed vagal stimulator, pacemaker, or spinal pain pump, which are not compatible with MRI.
7. Subjects must not have a history of seizures or neurologic conditions that may alter the structure of the brain.
8. Subjects must not be allergic to the metals used in electrodes for CES stimulation.
9. Subjects must not have a diagnosed autoimmune disease that better explains pain symptoms.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in Defense and Veterans Pain Rating Scale (DVPRS) from baseline | Baseline, 6 and 12 weeks post-intervention
  The Defense and Veterans Pain Rating Scale (DVPRS) is a pain assessment tool. Patients will rate their pain intensity on a scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain.
Change in Brief Pain Inventory (BPI) severity subscale from baseline | Baseline, 6 and 12 weeks post-intervention
  The BPI assesses pain severity and interference with function. The pain severity subscale consists of 4 items, each rated on a 0-10 numerical scale (0 = "no pain," 10 = "pain as bad as you can imagine"). Scores are averaged to yield a total range of 0-10. Lower scores reflect less severe pain and are considered favorable outcomes.
Change in Brief Pain Inventory (BPI) pain interference subscale from baseline | Baseline, 6 and 12 weeks post-intervention
  The pain interference subscale consists of 7 items rated on a 0-10 numerical scale (0 = "does not interfere," 10 = "completely interferes"), assessing the impact of pain on daily activities such as mood, walking ability, work, and enjoyment of life. Scores are averaged to create a total range of 0-10. Lower scores reflect less interference from pain and are considered favorable outcomes.

SECONDARY OUTCOMES:
Change in sit-to-stand/chair stand test | Baseline, 6 and 12 weeks post-intervention
  It involves repeatedly standing up and sitting down from a chair for a set period (30 seconds).
  The number of complete repetitions within the time limit is recorded.
Change in bicep(arm) curls | Baseline, 6 and 12 weeks post-intervention
  The test involves having the individual perform as many controlled arm curls as possible within a 30-second timeframe. The total number of controlled repetitions within the 30-second period is recorded.
Change in handgrip strength | Baseline, 6 and 12 weeks post-intervention
  Involves using a hand-held dynamometer to measure the maximum force exerted when squeezing the device. Maximun strength will be recorded.
Change in finger-tap test | Baseline, 6 and 12 weeks post-intervention
  The Finger Tapping Test (FTT) is a physical function assessment used to evaluate motor speed and coordination. It's a simple test where a person taps their index finger against their thumb as quickly as possible for a set period, often 10 seconds, and the number of taps is recorded.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS): sleep score | Baseline, 6 and 12 weeks post-intervention
  This measure focuses on the past seven days and assesses perceived difficulties with sleep onset, sleep continuity, and overall sleep quality.
  It includes a 5-point Likert scale (1=never to 5=always) for each item. Raw scores are summed, and then converted to T-scores, where 50 represents the average for the U.S. general population, and a standard deviation of 10. Higher T-scores represent better health.
Change in PROMIS: social isolation score | Baseline, 6 and 12 weeks post-intervention
  This measure focuses on the past seven days and assesses perceived difficulties with social isolation.
  The measure use a 5-point Likert scale (1=never to 5=always) for a total of 4 items item. Total possible score range from 4-20 with lower score correlating with better study outcome.
Change in PROMIS: alcohol use score | Baseline, 6 and 12 weeks post-intervention
  This measure focuses on the past seven days and assesses perceived difficulties with alcohol use.
  The measure use a 5-point Likert scale (1=never to 5=always) for a total of 37 items item. Total possible score range from 37-185 with lower score correlating with better study outcome.
Change in PROMIS: global health score | Baseline, 6 and 12 weeks post-intervention
  This measure focuses on the past seven days and assesses perceived difficulties with global health.
  The measure use a 5-point Likert scale (1=never to 5=always) for a total of 9 items item. Total possible score range from 9-45 with lower score correlating with better study outcome.
Change in PROMIS 29 score | Baseline, 6 and 12 weeks post-intervention
  PROMIS-29 involves assessing responses on a 1-5 scale (or 0-10 for pain intensity), then averaging responses within each of the seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) to create a raw score for that domain. These raw scores are transformed into T-scores, with a mean of 50 and a standard deviation of 10, to indicate health status relative to a reference population, where higher T-scores represent better health.
Change in SF-36 score from baseline | Baseline, 6 and 12 weeks post-intervention
  SF-36 is a multi-purpose, short-form health survey developed for assessing health-related quality of life. It measures eight health concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to personal or emotional problems, and mental health.
  Each scale score has a possible score range 0-100 scale, where 0 represents the worst possible health state and 100 represents the best.
  The scores for the items that contribute to each scale are averaged to produce a total score for the scale (possible range 0-100), higher score represents better outcome.
Change in Resting-State fMRI Connectivity measured with Seed-Based Functional Connectivity Analysis | Baseline, 6 and 12 weeks post-intervention
  This outcome assesses changes in functional connectivity within brain function networks relevant to chronic pathology through Pearson correlation between fMRI signal in relevant seed regions of interest. Higher FC within impaired brain function networks (e.g., fronto-temporal) and lower FC within abnormally enhanced (pain expression) represent better outcomes.
Change in Resting-State fMRI Connectivity measured with Independent Components Analysis | Baseline, 6 and 12 weeks post-intervention
  This outcome assesses changes in functional connectivity within the brain and between brain function networks relevant to chronic pathology. Independent Components Analysis (ICA) measures resting state network (IC) connectivity strength (expressed as z-sore) and between functional network connectivity (FNC). Higher IC strength within impaired brain function networks (e.g., fronto-temporal) and lower IC strength within abnormally enhanced (pain expression) represent better outcomes. Higher FNC in beneficent inter-network connections (e.g., between fronto-striatal and limbic networks) and lower FNC in malignant inter-network connections (e.g., default mode and pain expression networks) represent better outcomes.
Change in Magnetic Resonance Spectroscopy Metabolite: lactate | Baseline, 6 and 12 weeks post-intervention
  This outcome assesses changes in brain neurochemical composition across the study period.
  Magnetic Resonance Spectroscopy (MRS) will be used to measure water-scaled, tissue-corrected concentrations of lactate. Reductions in lactate represents better outcome.
Change in Magnetic Resonance Spectroscopy Metabolite: N-acetyl aspartate (NAA) | Baseline, 6 and 12 weeks post-intervention
  Magnetic Resonance Spectroscopy (MRS) will be used to measure water-scaled, tissue-corrected concentrations of N-acetyl aspartate (NAA). Reductions in NAA represents better outcome.
Change in Magnetic Resonance Spectroscopy Metabolite: choline | Baseline, 6 and 12 weeks post-intervention
  Magnetic Resonance Spectroscopy (MRS) will be used to measure water-scaled, tissue-corrected concentrations of choline. Reductions in choline represent better outcome.
Change in Magnetic Resonance Spectroscopy Metabolite: tCr | Baseline, 6 and 12 weeks post-intervention
  Magnetic Resonance Spectroscopy (MRS) will be used to measure water-scaled, tissue-corrected concentrations of total creatine (tCr). A decrease in tCr concentration, represents better outcome.
Change in Magnetic Resonance Spectroscopy Metabolites: Ratio of NAA/tCr | Baseline, 6 and 12 weeks post-intervention
  Ratio of NAA/tCr will also be quantified, as a decreased ratio of NAA/tCr has been linked to mitochondrial dysfunction in ill Gulf War Veterans. An increase in NAA/tCr ratio, represents better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Woodbury, MD, MSc, Principal Investigator — Emory University 404-727-8463; Lisa C Krishnamurthy, PhD, Principal Investigator — Emory University 404-712-5332
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Neuroimaging data (de-identified) will be shared for use in ENIGMA as part of the Chronic Pain Working Group Clinical outcomes (de-identified) for correlation with neuroimaging data Data may also be shared with the DOD and with other investigators
Supporting Information: Study Protocol, SAP
Time Frame: September 1, 2030-September 1, 2032
Access Criteria: - Data will be shared including with: DOD ENIGMA Chronic Pain Working Group Device manufacturer for the CES in case they would like to apply for an FDA indication
  - For the following type of analyses: Neuroimaging analysis Analysis of clinical outcomes
  - Through a data usage agreement